CLINICAL TRIAL: NCT01851486
Title: The Relationships Between the Noradrenergic, Opioid and Pain System
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Labortory focus was changed and study was not opened at all
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, d_yarnitsky, Professor, Head on Neurology Department, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 0393-12-RMB.CTIL
Record Dates: First submitted 2013-05-02; First posted 2013-05-10 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Experimental Pain Perception
MeSH Terms: interventions — Clonidine; Naloxone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Clonidine+ Saline (Active Comparator): Clonidine 0.15 mg and saline 0.15 mg/kg
  Interventions: Drug: Clonidine; Other: saline
- Clonidine + Naloxone (Active Comparator): Clonidine 0.15 mg and Naloxone 0.15 mg/kg
  Interventions: Drug: Clonidine; Drug: Naloxone
- Placebo +Naloxone (Active Comparator): Placebo 0.15 mg+ naloxone 0.15 mg/kg
  Interventions: Drug: Naloxone; Drug: placebo
- Placebo +saline (Placebo Comparator): Placebo 0.15 mg+ saline 0.15 mg/kg
  Interventions: Drug: placebo; Other: saline

INTERVENTIONS:
Drug: Clonidine — Clonidine 0.15 mg
  Arms: Clonidine + Naloxone; Clonidine+ Saline
Drug: Naloxone — naloxone 0.15 mg/kg
  Arms: Clonidine + Naloxone; Placebo +Naloxone
Drug: placebo
  Arms: Placebo +Naloxone; Placebo +saline
Other: saline
  Arms: Clonidine+ Saline; Placebo +saline

SUMMARY:
The role of alpha2 receptor agonist on pain perception and modulation will be examined. In addition whether this is mediated through the opioid system will be examined. Pain perception and modulation will be examined before and after administration of Clonidine or placebo together with Naloxone or saline.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Age 18-40
* No chronic disease

Exclusion Criteria:

* Subjects who suffer from chronic pain / pain syndrome
* use of anti-depressant or anti-psychotic drugs
* suffering from cardiovascular disease
* breast feeding

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The changes in pain responses after administration of alpha 2 agonist and mu receptor antagonist | 2 years
  The change in pain perception (pain thresholds and pain ratings of suprathresholds stimuli) and in the excitatory and inhibitory pain modulation responses (assessed by the temporal summation and conditioned pain modulation paradigms) will be examined before and after administration of alpha 2 agonist with and without mu receptor antagonist

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Health Care Campus, Haifa, Israel